CLINICAL TRIAL: NCT03004430
Title: Mantra Meditation as Adjunctive Therapy in Major Depression: a Randomized Controlled Trial
Brief Title: Mantra Meditation in Major Depression
Acronym: MAMED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: Diakonie Kliniken Zschadraß (Other)
Collaborators: University Hospital Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAMED001
Record Dates: First submitted 2016-12-14; First posted 2016-12-28 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Depression
Keywords: Mantra; Meditation
MeSH Terms: conditions — Depression | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MAM (Experimental): Mantra Meditation Group
  Interventions: Behavioral: Mantra Meditation
- PMR (Active Comparator): Progressive Muscle Relaxation Group
  Interventions: Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Mantra Meditation — Silent mantra meditation with spiritual mantra
  Arms: MAM
Behavioral: Progressive Muscle Relaxation — Progressive Muscle Relaxation
  Arms: PMR

SUMMARY:
To evaluate effects of mantra meditation on depressive symptoms if applied as adjunctive therapy to psychotherapy and/or antidepressant drugs and to explore if meditation leads to increased spirituality as a potential mediating factor of positive mental health.

DETAILED DESCRIPTION:
Primary objective To measure the difference in efficacy between treatment as usual (TAU) + Mantra meditation (MAM) 20min per day and TAU + progressive muscle relaxation (PMR) 20min per day in the treatment of depressive symptoms in patients with Major Depression after inpatient treatment, after 3 months and after 6 months of treatment as assessed by the Montgomery-Åsberg Depression Rating Scale (MADRS).

Secondary objectives (exploratory)

1. Differences between and within groups in self-rated depression, rumination, automatic negative thinking or trait-anxiety.
2. Differences between and within groups in measures of spirituality.
3. Correlation between measures of spirituality and change of psychometric scores.
4. Change in stress response and relaxation response after inpatient treatment, compared to baseline.
5. Difference in adherence and depth of practice between groups and within groups and correlation to psychometric outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients of open psychiatric ward
2. Written informed consent by patients who are competent to consent to study participation
3. Diagnosis of current episode of major depression as defined by DSM-IV criteria and diagnosed via structured interview (SKID) by a trained psychiatrist or psychologist. DSM-IV codes: 296.22, 296.23, 296.32, 296.33. Corresponding ICD-10 codes: F32.1, F32.2, F33.1, F33.2.
4. Male or female ≥18 years of age
5. BDI-II >= 20
6. Patients must be able to sit in a chair for at least 20 minutes
7. Patients live in the catchment area of the hospital

Exclusion Criteria:

Patients will be excluded for ANY ONE of the following reasons:

1. Any other current major psychiatric disorder is an exclusion criterion EXCEPT for the following:

   * Abuse of nicotine or dependence of nicotine;
   * Agoraphobia with or without Panic Disorder, Generalized Anxiety Disorder, Posttraumatic Stress Disorder, Specific Phobia, Social Phobia
   * Hypochondriasis, Pain Disorder, Somatization Disorder, Undifferentiated Somatoform Disorder
   * Sexual and Gender Identity Disorders
   * Eating disorders
2. Psychotic symptoms that are not compatible with diagnosis of unipolar depression
3. Acute suicidality
4. Diagnosis affecting cortisol levels such as type I diabetes mellitus, cancer, asthma, chronic hepatitis, chronic fatigue syndrome, or regular use of medications having an immuno-modulary effect (e.g. cytotoxic chemotherapy, corticosteroids, interferons);
5. Current practice of other forms of Mantra repetition such as the rosary, chanting, or Transcendental Meditation
6. Current participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
MADRS / SIGMA | 6 months
  The clinician-rated Montgomery and Asberg Depression Rating Scale (MADRS) [reproduced in the Appendix to this chapter] was developed in the late 1970s (Montgomery & Asberg, 1979) and this 10-item scale was designed to be sensitive to the effects of antidepressant medications, primarily tricyclic antidepressants. One of the original goals of the MADRS was to obtain an instrument that could be used by both psychiatrists and professionals without a specific or with minimal psychiatric training. From the original report of the MADRS, the inter-rater reliability ranged from 0.89 to 0.97. However, in a German study, significant differences resulted when the same patient was rated by various groups of caregivers (as described in Cusin, Yang, Yeung, & Fava, 2010). Hence, a structured interview guide (SIGMA) that has been developed for the MADRS (Williams, Kobak, & Montgomery, 2008) will be used in this study by trained psychologists exclusively.

SECONDARY OUTCOMES:
STAI-T | 6 months
  The State-Trait Anxiety Inventory (STAI) is an introspective psychological inventory consisting of 40 self-report items pertaining to anxiety affect. The STAI was constructed by Charles Spielberger, R.L. Gorsuch, and R.E. Lushene, based on the state-trait distinction proposed by Raymond Cattell in 1961. Their goal was to compile a set of items that could measure anxiety at both poles of the normal affect curve (state vs. trait). The STAI purports to measure one's conscious awareness at two extremes of anxiety affect, labeled state anxiety (A-state), and trait anxiety (A-trait), respectively. Affectivity ranges from immediate, transitory emotional states, through longer-lasting mood states, through dynamic motivational traits, ranging all the way up to relatively enduring personality traits. Higher STAI scores suggest higher levels of anxiety (C D Spielberger & Sydeman, 1994; Charles D Spielberger, 1987).
PTQ | 6 months
  The PTQ (Ehring et al., 2011) is a 15-item questionnaire assessing the tendency to engage in repetitive negative thinking independent of a disorder-specific content. Items are rated on a scale ranging from 0 (never) to 4 (almost always). The PTQ consists of three subscales: Core features of repetitive negative thinking, perceived unproductiveness of repetitive negative thinking , and repetitive negative thinking capturing mental capacity (sample item: 'My thoughts prevent me from focusing on other things'.). Confirmatory factor analysis provides support for a 3-factor solution. Assessment of the psychometric properties of the PTQ, including the Dutch version (Ehring, Raes, Weidacker, & Emmelkamp, 2012), has demonstrated high internal consistency (a = .93-.95), acceptable test-retest reliability (r = .69-.75), good convergent validity as well as good predictive validity in the prediction of symptom levels of anxiety and depression.
RSQ | 6 months
  The rumination scale of the Response Style Questionnaire (RSQ; Nolen-Hoeksema, 1991; German version: Kühner, Huffziger, & Nolen-Hoeksema, 2007) was used to assess repetitive negative thinking in the form of depressive rumination. The questionnaire consists of 22 items describing the individual's response to sad or depressed mood (e.g., "Think about how passive and unmotivated you feel") that are rated on a scale from '1' (never) to '4' (always). The RSQ is regarded as the standard measure of rumination; it has been used widely in clinical as well as non-clinical populations and has demonstrated high reliability and validity (Kühner et al., 2007, Luminet, 2004 and Nolen-Hoeksema, 2004).
ASP | 6 months
  Aspects of Spirituality (ASP) . The ASP questionnaire was developed to measure a wide variety of vital aspects of spirituality beyond conventional conceptual boundaries in secular societies. Both expert representatives of various spiritual orientations and also atheists were asked which aspects of spirituality are relevant to them (Büssing, 2006). Identified motifs we condensed to 40 items of the Aspects of Spirituality (ASP 1.0) questionnaire (7 factors; Cronbach ́s alpha = .94) (Büssing et al., 2007) which differentiates and quantifies cognitive, emotional, intentional and action-oriented matters of theism/belief, (esoteric) transcendence, existentialism, humanism etc. The reliable and valid instrument is suited to be used in health care research (Büssing et al. 2007).
SpREUK | 6 months
  The SpREUK was developed to investigate whether or not patients with chronic diseases living in secular societies rely on spirituality as a resource to cope with illness. The SpREUK questionnaire relies on essential motifs found in counseling interviews with chronic disease patients (i.e., having trust/faith; search for a transcendent source to rely on; reflection of life and subsequent change of life and behavior). The instrument is suited to be used in health care research (A Büssing, Ostermann, & Matthiessen, 2005).
EEQ | 6 months
  A new instrument for the measurement of exceptional experiences, which considers both frequency and individual evaluation of exceptional experiences. A principal component factor analysis extracted four factors (positive spiritual experiences, experiences of deconstruction/ ego loss, psychopathological experiences and dream-type experiences), which explain 49% of the variance. The 25-item short form of the instrument shows good psychometric properties (range for Cronbach's alpha: r = 0.67-0.89, range for test- retest reliability after 6 months r = 0.66-0.87). The instrument shows adequate discriminant and convergent validity (Sense of Coherence, Social Support, Mental Distress and Transpersonal Trust) and can discriminate between spiritual practising and non practising individuals (Kohls & Walach, 2006).
ICPH | 6 months
  Specific mind-body-interventions (i.e., yoga, quigong, therapeutic eurythmy, mindfulness-based meditation etc.) require an active (emotional) engagement of individuals practicing it. Apart from direct physiological effects, an active emotional engagement seems to be important. This type of engagement can be conceptualized as an 'inner involvement ́ (Büssing et al. 2011). Lacking this attitude in terms of an inner resistance towards the practices may lead to reduced engagement, adherence, and thus treatment efficacy. The ICPH scale ("Inner Correspondence / Peaceful Harmony with Practices") was developed to measure this 'inner correspondence in clinical studies addressing the efficacy of mind body practices involving physical movements. While it is suitable for progressive muscle relaxation, wording needs to be adjusted for mantra meditation (Arndt Büssing, Edelhuser, Weisskircher, Fouladbakhsh, & Heusser, 2011).
HRV | 1 month
  Change of Cardiovagal Index (CVI), a normalized measure of heart rate variability (HRV), in stress response and relaxation response after inpatient treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Holger C Bringmann, Dr. med., Principal Investigator — Diakoniekliniken Zschadraß
Locations (1):
- Diakoniekliniken Zschadraß, Colditz, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ospina MB, Bond K, Karkhaneh M, Tjosvold L, Vandermeer B, Liang Y, Bialy L, Hooton N, Buscemi N, Dryden DM, Klassen TP. Meditation practices for health: state of the research. Evid Rep Technol Assess (Full Rep). 2007 Jun;(155):1-263. PMID 17764203
- [Result] Ospina MB, Bond K, Karkhaneh M, Buscemi N, Dryden DM, Barnes V, Carlson LE, Dusek JA, Shannahoff-Khalsa D. Clinical trials of meditation practices in health care: characteristics and quality. J Altern Complement Med. 2008 Dec;14(10):1199-213. doi: 10.1089/acm.2008.0307. PMID 19123875
- [Result] Goyal M, Bass EB, Haythornthwaite JA. Meditation intervention reviews--reply. JAMA Intern Med. 2014 Jul;174(7):1195. doi: 10.1001/jamainternmed.2014.1393. No abstract available. PMID 25003880